CLINICAL TRIAL: NCT02844569
Title: A Volumetric Analysis of Soft and Hard Tissue Healing for Ridge Preservation and Socket Seal After Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0832
Record Dates: First submitted 2016-07-21; First posted 2016-07-26 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2018-11

CONDITIONS: Tooth Extraction
Keywords: Dental Implants; Bone Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Extraction treated with xenograft bone substitute (BioOss Collagen®) + 3D-collagen matrix (Mucograft Seal®).
  Interventions: Device: Xenograft bone substitute; Device: 3D-collagen matrix
- Control (Active Comparator): Extraction treated with xenograft bone substitute (BioOss Collagen®) + collagen dressing (HeliPlug®).
  Interventions: Device: Xenograft bone substitute; Device: Collagen dressing

INTERVENTIONS:
Device: Xenograft bone substitute — Subjects requiring tooth extraction will have the hopeless tooth extracted. The extraction socket will be treated with xenograft bone substitute. At 6 months post-extraction a dental implant will be placed at the extraction site.
  Other Names: BioOss Collagen®
Device: Collagen dressing — Subjects requiring tooth extraction will have the hopeless tooth extracted. The extraction socket treated with xenograft bone substitute will receive a collagen dressing to cover the surgical site.
  Other Names: HeliPlug®
  Arms: Control
Device: 3D-collagen matrix — Subjects requiring tooth extraction will have the hopeless tooth extracted. The extraction socket treated with xenograft bone substitute will receive a 3D collagen matrix to cover the surgical site.
  Other Names: Mucograft Seal®
  Arms: Test

SUMMARY:
This study will be a randomized clinical trial involving a total of 24 subjects. The investigators propose to recruit subjects into 2 groups: 1) Extraction treated with xenograft bone substitute (BioOss Collagen®) + collagen dressing (HeliPlug®), 2) Extraction treated with xenograft bone substitute (BioOss Collagen®) + 3D-collagen matrix (Mucograft Seal®). All subjects recruited will have already been approved and treatment planned for extraction + implant placement by non-study personnel to avoid any potential conflict of interest. All subjects will have radiographs that show the tooth planned for extraction. Each subject will be eligible for only 1 tooth extraction + dental implant rehabilitation. After tooth extraction, subjects will receive a standard site preservation therapy consisted with xenograft bone substitute + collagen dressing or the alternative site preservation therapy consisted with xenograft bone substitute + 3D-collagen matrix. After the conventional 6-month healing period, subjects will receive a dental implant in the previous extracted site. During the dental implant procedure, a 2x5mm bone core biopsy + a 2mm gingival biopsy will be obtained from the implant site. Biopsy samples will be stored for future histological and histochemical analysis. After dental implant placement, all subjects will receive a healing abutment for soft tissue healing prior to implant restoration.

During the 6-month healing time after tooth extraction and site preservation therapy, subjects will return at week-1, week-2, week-4, month-3, and month-6 for intra-oral scanning for soft tissue volumetric acquirement. Subjects will receive a Cone beam computed tomography (CBCT) prior to extraction for the baseline hard-tissue volume measurement and appropriate extraction planning and at 6-month post-extraction for volumetric measurement and appropriate implant treatment planning.

Hard tissue analysis will be performed to compare linear ridge remodeling (baseline vs. 6-month healing). CBCT images will be analyzed by non-contact reverse engineering system. Soft tissue volumetric analysis will be performed to compare the soft tissue healing between BioOss Collagen + Mucograft Seal and BioOss Collagen + Collagen Dressing. Images captured with an intra-oral scanner collected at baseline, week-1, -2, -4, month-3, and month-6.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adult males or females age 18 to 80 years (inclusive).
* Subjects must be able and willing to follow study procedures and instructions in English.
* Subjects must have read, understood and signed an informed consent form in English.
* Subjects must have a maxillary premolar, canine, lateral incisor, or central incisor with a restorative or periodontal hopeless prognosis (Kwok and Caton 2007), in which an implant is indicated without any sinus lift required.
* Subjects undergoing implant placement should be in adequate periodontal health prior to implant placement. This includes having probing depth ≤ 4 mm for all remaining teeth at the same quadrant of the proposed implant placement. Patients with periodontal probing sites with probing depths of up to 5 mm may also be included if bleeding on probing in these sites is absent. Each subject should be considered to be periodontally stable prior to the implant surgery.

Exclusion Criteria:

* Individuals who have a chronic disease with oral manifestations.
* Individuals who exhibit gross oral pathology.
* The use of either antibiotics or chronic use (more than 7 days) of NSAIDs within 1 month prior to screening examination.
* Individuals that require antibiotic prophylaxis prior to dental treatment.
* Chronic treatment (i.e. two weeks or more) with any medication known to affect periodontal status (e.g. phenytoin, calcium antagonists, cyclosporine, Coumadin) within 1 month prior to screening examination.
* Uncontrolled diabetes mellitus (HbA1c >7) within 3 months prior to screening examination.
* Individual with uncontrolled parafunctional habits, such as clenching and bruxing on objects, that could adversely impact implant survival.
* Individuals with a history of intravenous bisphosphonates.
* Individuals with active infectious diseases such as hepatitis, HIV or tuberculosis.
* Current cigarette smokers.
* Individuals who are known to be pregnant, breastfeeding or planning to become pregnant within 6 months.
* Individuals with blood disorders (hemophilia) and /or currently taking anticoagulant medications, such as heparin, warfarin, or clopidogrel.
* Individuals receiving any therapy known to affect healing, such as high dose corticosteroids, radiation therapy or chemotherapy.
* Individuals allergic to topical or local anesthesia.
* Individuals who require maxillary sinus augmentation prior to dental implant therapy.
* Individuals with dehisced, fenestrated, or fractured labial/buccal alveolar bone plate determined after baseline CBCT or after tooth extraction where more than 50% of the buccal bone height is not present. In this case, if the surgeon determines that guided bone regeneration (bone graft and membrane) is needed to repair the defect, it will be done at no cost to the subject, but the subject will be excluded from the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Marchesan, DDS, PhD, Principal Investigator — Assistant Professor Periodontology
Locations (1):
- General & Oral Health Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9-36 months following publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 9-36 months following publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test | Control
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Full Range); unit: years] | 45.2 [31 to 60] | 56.4 [38 to 69] | 50.8 [31 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Buccal Plate Thickness From Baseline to Month 6
Description: The thickness difference between baseline and 6 months will be measured by the difference in mm using cone-beam computed tomography.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test | Control
Number analyzed (Participants) | 10 | 8
mm | 1.85 (0.72) | 1.25 (0.45)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Superiority; p = 0.11, t-test, 2 sided

2. Primary Outcome: Change in Buccal Soft Tissue Volume Between Baseline and 6 Months
Description: The soft tissue volume change between baseline and 6 months based on 3D images captured with intra-oral digital scanner.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Test | Control
Number analyzed (Participants) | 12 | 12
mm^3 | 68.6 (25.4) | 87.6 (39.1)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Superiority; p < 0.01, Mixed Models Analysis

3. Primary Outcome: Change in Buccal Bone Volume Between Baseline and 6 Months
Description: The buccal bone volume change between baseline and 6 months will be calculated from cone-beam computed tomography data.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Test | Control
Number analyzed (Participants) | 12 | 12
mm^3 | 72.6 (30.7) | 60.9 (37.3)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Superiority; p = 0.66, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From time of extraction through 7 months after extraction
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT02844569/Prot_SAP_000.pdf